CLINICAL TRIAL: NCT05675293
Title: Effectiveness of Iontophoresis in Managing Uterine Cervicitis
Brief Title: Cervicitis by Iontophoresis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, MARIAM HELMY, Practitioner, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IONTOPHORESIS FOR CERVICITIS
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: CERVICITIS
MeSH Terms: conditions — Uterine Cervicitis | interventions — Iontophoresis; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL ARM (Experimental)
  Interventions: Device: IONTOPHORESIS
- CONTROL ARM (Active Comparator)
  Interventions: Drug: ORAL ANTIBIOTIC

INTERVENTIONS:
Device: IONTOPHORESIS — The process of increasing the penetration of drugs into the skin by application of an electric current
  Arms: EXPERIMENTAL ARM
Drug: ORAL ANTIBIOTIC — Oral Antibiotic
  Arms: CONTROL ARM

SUMMARY:
The purpose of the study is to:

Investigate effect of iontophoresis on managing uterine cervicitis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients have vaginal discharge.
2. All patients have irregular vaginal bleeding, especially after sexual intercourse.
3. All patients have dyspareunia.
4. All patients have Lower abdominal pain.
5. Group A: 20 women will receive oral medication (antibiotic zesrosin) and hot water with antiseptic.
6. Group B: 20 women will receive medication by iontophoresis (antibiotic ceftriaxone) and hot water with antiseptic.

Exclusion Criteria:

1. Patients with a history of hypersensitivity or adverse reactions associated with the delivered drug in (ceftriaxone).
2. Patients with prior medical histories of cardiac arrhythmias or hypercoagulability should not receive the procedure near cardiac pacemakers and superficial blood vessels.
3. In the vicinity of embedded wires, stapes, orthopedic implants, and areas of skin with lesions and impaired sensation.
4. It either should not be used or used with extreme caution during pregnancy.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Difference in change in Urine Analysis and Cervical swab results in both groups | 7 Days difference between pre and post tests
  Presence of Pus Cells in Urine Analysis and a Positive Cervical swab results